CLINICAL TRIAL: NCT05920733
Title: Healthy Lifetime - Sustainability and Quality Study - PHASE 2
Brief Title: Healthy Lifetime - Phase 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Kathleen Potempa, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00223787
Record Dates: First submitted 2023-05-18; First posted 2023-06-27 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Aging Well
Keywords: nurse coaching; motivational interviewing; aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HealthyLifetime Group (Experimental): This project is designed to prepare and equip the participant for improved self-care capacity, motivational insight, health-related problem solving and decision-making.
  Interventions: Behavioral: Nurse-led health coaching

INTERVENTIONS:
Behavioral: Nurse-led health coaching — This project is an 6-month program providing an initial 2-month intensive evaluation and personalized virtual individual health coaching experience that is designed to prepare and equip the participant for improved self-care capacity, motivational insight, health-related problem solving and decision-making. This intensive period will then be followed by monthly 30-minute Nurse Coach assessment and individual coaching 'check-in' virtual visits, continued use of the electronic platform tools and health tracking system, and access to group 'virtual coaching' on tailored topics of interest to the cohort.
  Other Names: HealthyLifetime

SUMMARY:
HealthyLifetime (HL) is a person-centered program that enables older adults to maximize health and optimize functioning - the necessary requisite to successfully remaining independent in their preferred home setting as long as possible, i.e., to age in place.

DETAILED DESCRIPTION:
HL seeks to intervene early in the aging process when individuals have the best chance for longer term benefits of changing their health behavior, as a means to stave off functional decline, and minimize the onset or exacerbation of chronic conditions. And, for individuals who are experiencing any of the barriers described above, our HL program's Nurse Coaches are prepared and experienced in helping them achieve their highest level of functioning and self-care capacity, while integrating and collaborating with, but not duplicating, their medical services such as primary care, specialty care, and case management or medical social services. While the latter medically oriented services support clinical management, they do not focus on helping older adults maximize health and function by building self-care capacity, long term health behavior change capacity and the functional resilience necessary to sustain or regain independent living.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read, speak English and hear - but may use glasses or hearing aids, if needed;
* Be able to tell us their age, their date of birth, address, and phone number, as well as write down and explain their health problems;
* Have their own computer or iPad (Tablet) with an Internet connection, a working camera and microphone. and
* Be able to use their computer/tablet to connect to video chat sessions like Zoom in a private space in their home or a private room.

Exclusion Criteria:

* People who, in the last month, have used the Emergency Room (ER) or stayed in the hospital.
* Are not verified users of Medicaid Home Help services [we will check with the Michigan Department of Health and Human Service to verify that you receive these services using your name, date of birth, and Medicaid identification number];
* Have a new major health problem that they are seeing a doctor about more than once per month;
* Have been told their illness is not curable;
* Cannot remember their name, date of birth or their health problems;
* Cannot use glasses or a hearing aid to see or hear well enough to read materials on the computer or talk to the nurse easily; and,
* Do not have, or cannot use, a computer, iPad or other device with the Internet at home to use Zoom (e.g., internet streaming).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Participant Self- rated health score | At 0, 8 and 20 weeks after study enrollment.
  Participants perception of their health on a scale of 1= Excellent to 5 = Poor
Change in Self-efficacy in ability to continue essential life activities score | At 0, 8 and 20 weeks after study enrollment.
  Confidence of the participant in doing certain activities on a scale of 1= Not at all confident to 10 = Totally Confident. For the purposes of answering these questions, confidence is defined as the belief in the participant's chances of being able to do and/or complete an activity (e.g., hobbies and recreation, social visits, chores, errands, etc.) or task (e.g., hobbies and recreation, social visits, chores, errands, etc.) successfully however the participant defines it.
Change in Independent self-care agency score | At 0, 8 and 20 weeks after study enrollment.
  Confidence in doing certain activities, e.g., stick to behavior changes, meet goals, and improve health, on a scale of 1= Not at all confident to 10 = Totally Confident
Change in Health Habits score | At 0, 8 and 20 weeks after study enrollment.
  Activities that participants engage in that affect health in a negative or positive way, e.g., smoking (yes or no), alcohol (number of drinks per week), exercise (0 = none to 4= more than 3 hours/week), food choices (seldom or never to 2 or more times a day)
Change in Goal attainment score | At 0, 8 and 20 weeks after study enrollment.
  Health goals (up to 3) of participants and importance of goal (1= Not at all important now to 10 = highest importance now) and confidence in achieving goal (1= Not confident at all to 10 = Completely Confident)
Change in Quality of Life score | At 0, 8 and 20 weeks after study enrollment.
  Questions about how participant experiences their quality of life. Covers six areas and includes how satisfied they are with these areas, and how important they are to them.
  Uses a scale where "0" = "Do not agree at all" and "4" = "Agree completely"
Change in Lifestyle Habits | At 0, 8 and 20 weeks after study enrollment.
  Questions about tobacco and alcohol use: Do participants use alcohol and/or tobacco, and, if so, how much
Change in Food Consumption | At 0, 8 and 20 weeks after study enrollment.
  Participants report how frequently they eat foods from different food groups, e.g., vegetables, fruits, grains, dairy, sugary, etc.
Change in Exercise and Activities | At 0, 8 and 20 weeks after study enrollment.
  DURING THE PAST 7 DAYS, even if it was not a typical week for participants, how much total time (for the entire week) did they spend on each of various exercises or activities, e.g., walking, swimming, bicycling, etc.
Change in Vigorous Activity | At 0, 8 and 20 weeks after study enrollment.
  Number of days out of the past seven did participants do vigorous or moderate activities at work, as part of their house and yard work, to get from place to place, and in their spare time for recreation, exercise, or sport.
Change in Level of independence in household activities score | At 0, 8 and 20 weeks after study enrollment.
  Ability to do daily living activities such as shopping, cooking, managing medications, etc. on a scale where 1 = Not at all Confident to 10 = Totally Confident
Change in Health Impact | At 0, 8 and 20 weeks after study enrollment.
  Using a "1" to "10" scale where "1" = "Almost never" and "10" = "Almost totally", participant selects ONE number which best represents how much their health impacts their ability to do or participate in an activity AT THE PRESENT TIME.
Change in Confidence in ability to manage symptoms score | At 0, 8 and 20 weeks after study enrollment.
  How confident the is participant that they can keep health symptoms/problems from interfering with the things they want to do, e.g., fatigue, physical discomfort, emotional distress, etc. on a scale where 1 = Not at all Confident to 10 = Totally Confident
Change in Level of Symptomatology score | At 0, 8 and 20 weeks after study enrollment.
  Frequency with which participants experience symptoms such as physical discomfort, pain, fatigue, etc. on a scale where 0 = Never to 5 = Always
Change in Other Symptoms | At 0, 8 and 20 weeks after study enrollment.
  Questions ask how often a participant is bothered by psychological and emotional symptoms such as feeling nervous, worry, anxiety, sadness, etc. On a scale from 0 Not at All to 3 Nearly Every Day.

SECONDARY OUTCOMES:
Higher values of primary measures at 8 weeks: persistence at 20 weeks | 20 weeks after study enrollment
  Are effects of program noted at 8 weeks still present at 20 weeks.
Change in Self-reported medical visits | At 0, 8 and 20 weeks after study enrollment.
  Number of unplanned medical visits with doctor or primary medical provider in past 2 months (0/none to 10), emergency room visits (0/none to10), overnight stay in hospital (0\none to 10).
Change in Social Network and Support score | At 0, 8 and 20 weeks after study enrollment.
  Number of friends and relatives participants interact with/rely on. Scale from None to Nine or more.
Change in type and source of At-home Support | At 0, 8 and 20 weeks after study enrollment.
  Do the type (healthcare, chores, meals, etc) and source (Medicare, Medicaid, other insurance, etc.) of help received by participants indicated in answers to survey questions change over course of study.

OTHER OUTCOMES:
Change in Perception of health now and in 3 years score | At 0, 8 and 20 weeks after study enrollment.
  Participant thinks health now is and in three years will be 1 = Excellent to 5 = Poor.
Change in Medication taking self care efficacy score | At 0, 8 and 20 weeks after study enrollment.
  Confidence of participants (on a scale where 0 = Not at all Confident to 2 = very Confident) in taking their medications correctly under different conditions, e.g., if take several medication each day, are away from home, if cause side effects, etc.
Health Conditions | At 0, 8 and 20 weeks after study enrollment.
  Participants are asked whether a medical provider may have told them that they have one or more common health problems, e.g., heart disease, high blood pressure, diabetes, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Potempa, PhD, Study Director — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No